CLINICAL TRIAL: NCT06953167
Title: Cognitive Health in Ageing Register: Investigational and Observational Trial Studies in Dementia Research (CHARIOT): Prospective Readiness Cohort (PRO) Longitudinal Study
Acronym: CPLS
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE ID: 174407; IRAS: 339745 (Other: IRAS)
Record Dates: First submitted 2025-04-03; First posted 2025-05-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease (AD)
Keywords: Alzheimer's disease; Dementia; Longitudinal Study; Biomarkers; CHARIOT-PRO; Amyloid; Cognition; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 825 participants who underwent CPSS1 screening have already had a Genome Wide Association Scan (GWAS) and APOE genotyping. A DNA sample for GWAS and APOE genotyping will be collected during the CPLS Study Entry Visit from all potential participants and GWAS will be performed in all cases of missing genetic data. The aim will be to evaluate the role of APOE status individually and of the polygenic risk score (PRS) in risk assessment of cognitive differing cognitive and ATN biomarker trajectories.
  Urine, blood (including for serum and plasma) and saliva samples will be collected and stored to allow for the future investigation of biomarkers associated with AD, through targeted or untargeted (omics) assays. Optional faecal samples will be collected for studies of the gut microbiome and its relationship to AD.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals who previously completed CHARIOT:PRO Substudy (CPSS1) screening.: All individuals who completed CPSS1 screening are well-characterised adults now aged >65 years old, with documented measurement of amyloid load and a global CDR score of 0 at the time of CPSS1 screening (2015-2018). They completed all CPSS1 screening assessments including the PACC and RBANS cognitive batteries, physical and neurological evaluation, clinical laboratory tests, quantitative and functional brain MRI studies, and (based on personal choice), either a PET scan or CSF collection via LP.
  The current project seeks to extend follow-up of CPSS1 study participants for at least another three years. Because CPSS1 screening began in 2015, this three-year follow-up will result in a total follow-up period of up to 12 years from CPSS1 screening for some participants.

SUMMARY:
Alzheimer's disease is a degenerative condition affecting the brain and is the most frequent form of dementia in older adults. Dementia is currently a major healthcare issue in the UK, affecting approximately a million people. The progression of the disease varies between individuals and the early stages may be characterised by only minimal changes in memory and thinking. These changes could remain undetected as the symptoms may be mistakenly regarded as normal age-related forgetfulness. However, dementia is not part of the normal ageing process.

The disease process is now known to start at least 20 years prior to the emergence of symptoms. A protein called amyloid starts to deposit in the brain, forming clumps referred to as 'plaques'. Another protein called tau sticks to other tau molecules inside the brain cell and forms structures called 'tangles'. These changes cause damage to the brain cells, disrupting their normal functioning, leading to inflammation and ultimately destruction of the brain cells.

So far, there is no cure for Alzheimer's disease, but by better understanding the changes that occur over time in the brain, scientists can find ways of detecting and therefore diagnosing and treating the disease earlier. One way in which scientists learn about how a disease develops, is by following people unaffected by the condition over an extended period of time. The same tests and sample collections are repeated to monitor any clinical changes. These are known as longitudinal studies, and CHARIOT:PRO studies are examples of this.

The CHARIOT:PRO Longitudinal Study (CPLS) is an observational study of 600 participants aged >65 years old which aims to evaluate cognition (thinking abilities) and biomarkers (biological markers which indicate the presence of disease e.g. amyloid) over time in older adults. The participants in CPLS were all screened as part of the CHARIOT:PRO Sub-Study (CPSS1) in 2015-2017.

Visit 1 will be conducted within eight weeks after the Study Entry Visit (SEV). Visits 2-7 will follow at six-monthly intervals from Visit 1. During visits, information relating to health, medication, family history of dementia, self-reported cognitive function and anthropometrics will be collected. The cognitive assessments PACC5 and RBANS will be administered along with a measure of executive function (Trail Making Test). Participants will be provided with self-reported questionnaires to be completed at each onsite visit. Blood samples will be taken once a year i.e. Month 0, 12, 24 and 36.

The purpose of CPLS is to continue to build on the vital data and samples already kindly donated by participants screened for CPSS1. This will provide valuable information that will enhance understanding of the earliest stages of Alzheimer's disease before obvious symptoms start to appear. Importantly, the Investigators hope to identify predictive markers of disease, which will help doctors to select the right drugs, and develop other approaches like lifestyle guidance to prevent or delay Alzheimer's disease in the future.

This study is sponsored by Imperial College London, led by the Principal Investigator Professor Lefkos Middleton and is funded by Gates Ventures.

DETAILED DESCRIPTION:
The aim of the study is to prospectively evaluate factors and markers associated with varying cognitive performance and longitudinal trajectories in individuals with differing levels of brain amyloid burden cross-sectionally as defined by PET imaging or Aβ42 CSF measurements (at CPSS1 screening), over a period of up to 12 years from CPSS1 screening.

Two C2N assays, i.e. the plasma Precivity AD2 and Multi-Tau assays, will be used at baseline and end -of-study, to assess the amyloid and tau cerebral burden, shown to have a comparable performance to PET and CSF. The former simultaneously quantifies specific plasma amyloid beta and tau peptide concentrations to calculate the Aβ42/40 Ratio and p-tau217/np-tau217(p-tau217 Ratio). The ratios are combined into a proprietary statistical algorithm to calculate the Amyloid Probability Score 2 (APS2), a numerical value ranging from 0-100, that determines whether a patient is Positive (has high likelihood) or Negative (has low likelihood) for the presence of abnormally high brain amyloid plaques by amyloid PET scan.A negative (0 - 47) is consistent with a negative amyloid PET scan; it reflects a low likelihood of brain amyloid plaques and is therefore not consistent with a neuropathological diagnosis of Alzheimer's disease (AD). A positive (48 - 100) is consistent with a positive amyloid PET scan; it reflects a high likelihood of brain amyloid plaques, one of the neuropathological findings of Alzheimer's disease (AD).

The Multi-Tau assay measures the individual values and rations of phosphorylated and non- phosphorylated p/non p-tau 217, p/non p-t181 and p/non p- t205. The presence of high amyloid and/or tau cerebral burden alone does not establish a clinical diagnosis of AD and the APS2 and multi-tau results will be interpreted in conjunction with other patient information and will be clinically correlated.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants must meet all inclusion criteria for the study, as follows:

  1. Male or Female, aged >65years
  2. Willing and having capacity (as assessed according to MCA 2005) to provide written informed consent and to participate in the study, OR (if lacking capacity) has a nominated consultee (as described in the MCA 2005 and Chapter 11 of the MCA Code of Practice 2007) who is able to advise that this is what the participant would have wished.
  3. Have completed CPSS1 amyloid screening using either amyloid PET scanning or CSF Aβ42 measurement.
  4. Be fluent in and able to read and write in English and have adequate hearing and visual acuity to complete the required psychometric tests.
  5. Be willing and able to adhere to the study visits and assessments specified in this protocol, and the reasonable requests and expectations of the study staff.
  6. Have a reliable informant - study partner (relative, partner, or friend) who is willing to provide their informed consent to participate, as a source of information. The study partner must be over 18 years old and should be fluent in and able to read and write in English. The informant must have sufficient contact with the participant and sufficient cognitive ability such that the Investigator feels that they can provide meaningful information about the participant's daily functioning. At a minimum, they must be in contact with the participant at least twice per month (in person, via telephone or other audio/visual communication). The study partner will be required in-person at the V1 visit. However, they can complete all subsequent visits remotely, or in-person if required.

Exclusion Criteria:

* To be eligible, participants must not meet any of the exclusion criteria for the study, as follows:

  1. Participant has any disability that would prevent completion of study procedures or assessments (e.g. blindness or significant visual impairment, deafness or significant hearing impairment, speech impairment, or sensory or motor dysfunction), or has any condition or situation/circumstance for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g. compromise the participant's well-being), or that could prevent, limit, or confound the results of protocol-specified assessments and cognitive testing.
  2. Unable to comply with the study-specific requirements.
  3. History of alcohol or drug dependence or abuse, as defined by the most current version of the DSM criteria within the last 3 years.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Well characterised cohort of participants who had completed all clinical, cognitive, biochemical and imaging screening assessments (during 2015-2018) required for study entry into CPSS1; were then >60 years old, with documented evidence of amyloid status and were, then, cognitively unimpaired.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Index scores | 8.5 years
  Raw scores are tallied for each of the 12 subtests and converted into five cognitive domain-specific Index scores (Immediate Memory, Delayed Memory, Language, Attention, Visuospatial Construction). Each Index score has a mean of 100 and an SD of 15, with a range of 40 to 160. Higher RBANS Index scores indicate better cognitive performance.
Change from baseline in the Preclinical Alzheimer Cognitive Composite (PACC) component scores | 8.5 years
  The raw score ranges for each test are as follows: Mini-Mental State Examination (MMSE): 0-30; Logical Memory (Wechsler Memory Scale) - Immediate Recall: 0-25; Delayed Recall: 0-25; Digit Symbol Substitution Test (DSST): 0-93; Free and Cued Selective Reminding Test (FCSRT) - Immediate Recall: 0-48 and Delayed Recall: 0-16; and Category Fluency (alternatively known as semantic fluency): 0-40. Across all PACC components, higher scores indicate better cognitive performance.

SECONDARY OUTCOMES:
Change from baseline in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Scale Score | 8.5 years
  RBANS raw scores are initially tallied for each of the 12 subtests and then converted into Index scores. These combined scores are further converted into a Total Scale Score, adjusted for age. The Total Scale Score is represented as a composite t-score with a mean of 100, a standard deviation (SD) of 15, and a range of 40-160. Higher RBANS Total scores indicate better cognitive performance.
Change from baseline in the Preclinical Alzheimer Cognitive Composite (PACC) composite score | 8.5 years
  Each component score will be transformed into a z-score. These z-scores will then be summed to form the PACC composite score. There is no fixed minimum or maximum for z-scores: a z-score of 0 represents average performance compared to a reference group; a negative z-score indicates below-average performance; and a positive z-score indicates above-average performance. Higher PACC composite scores indicate better cognitive performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom